CLINICAL TRIAL: NCT01978015
Title: Blood-aqueous Barrier Changes After the Use of Timolol and Prostaglandin Analogues Fixed Combination in Pseudophakic Patients With Primary Open Angle Glaucoma
Brief Title: Blood-aqueous Barrier Changes After the Use of Timolol and Prostaglandin Analogues Fixed Combination in Pseudophakic Patients With POAG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Alana Mendonça de Santana, Santana AM, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP424/2010; CAAE0319014600010 (Other: CAAE0319014600010)
Record Dates: First submitted 2013-10-25; First posted 2013-11-07 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-10

CONDITIONS: Uveitis, Anterior; Cystoid Macular Edema
Keywords: primary open angle glaucoma; timolol; prostaglandin analogues
MeSH Terms: conditions — Uveitis, Anterior; Macular Edema; Glaucoma, Open-Angle | interventions — Travoprost; Latanoprost; Xalacom; Bimatoprost; Ganfort; Dextrans; Hypromellose Derivatives

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- latanoprost and timolol maleate fixed combination (Experimental): Latanoprost 0.005% and timolol maleate 0,5% fixed combination was dropped once daily at 8 p.m. for 6 months
  Interventions: Drug: latanoprost and maleate timolol fixed combination
- bimatoprost and timolol maleate fixed combination (Experimental): bimatoprost 0.03% and timolol maleate 0,5% fixed combination was dropped once daily at 8 p.m. for 6 months
  Interventions: Drug: bimatoprost and timolol maleate fixed combination
- dextran and hypromellose (Placebo Comparator): A control group of patients with POAG and pseudophakic after trabeculectomy without medication. These patients received a lubricant drop twice daily at 8 a.m. and 8 p.m. for 6 months
  Interventions: Drug: dextran and hypromellose
- travoprost and timolol maleate fixed combination (Experimental): Travoprost 0.004% and timolol maleate 0,5% fixed combination was dropped once daily at 8 p.m. for 6 months
  Interventions: Drug: travoprost and timolol maleate fixed combination

INTERVENTIONS:
Drug: travoprost and timolol maleate fixed combination — travoprost 0.004% and timolol maleate 0,5%, 1 eye drop at 8p.m. for 6 months
  Other Names: Duo-travatan
  Arms: travoprost and timolol maleate fixed combination
Drug: latanoprost and maleate timolol fixed combination — Latanoprost 0.005% and timolol maleate 0,5%, 1 eye drop at 8 p.m for 6 months
  Other Names: Xalacom
  Arms: latanoprost and timolol maleate fixed combination
Drug: bimatoprost and timolol maleate fixed combination — bimatoprost0.03% and timolol maleate 0,5%, 1 eye drop at 8 p.m for 6 months
  Other Names: Ganfort
  Arms: bimatoprost and timolol maleate fixed combination
Drug: dextran and hypromellose — Dextran 70 and hypromellose, lubricant eye drop at 8 a.m and 8 p.m for 6 months
  Other Names: Lacribell
  Arms: dextran and hypromellose

SUMMARY:
Glaucoma, a progressive optic disc neuropathy causing visual field reduction, is the second leading cause of world blindness. The treatment of glaucoma is mainly based in reducing intraocular pressure (IOP) with topical medications. Many patients required two or more medications to achieve a target IOP. Combinations of B-blockers and prostaglandin analogs (PGA) are frequently used in clinical practice because their additive effect in lowering IOP levels. The aim of this study was to investigate the effects of fixed combinations of timolol maleate and PGA on the blood-aqueous barrier and evaluate the measurement of foveal thickness in pseudophakic patients with primary open-angle glaucoma (POAG).

DETAILED DESCRIPTION:
Most studies found a lower incidence of systemic and ocular adverse events with fixed combinations than with the unfixed combinations. Fixed combinations are better tolerated than their respective prostaglandin analogue. However, among the most serious side effects induced by PGA are the breaking down of the blood-aqueous barrier (BAB) and the development of cystoids macular edema (CME). Also, timolol maleate drops increase protein concentration in the human and benzalkonium chloride, eye drops preservative induces anterior chamber inflammation. This randomized, masked-observer, prospective clinical trial was approved by the Ethics Committee of the University of Campinas, and it adhered to the tenets of the Declaration Of Helsinki. Written informed consent was obtained from each patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible for participation if they met the following inclusion criteria: age older than 18 years, pseudophakia and diagnosis of primary open angle glaucoma (an untreated IOP levels of more then 21 mmHg, specific changes in the optic disc or specific visual fields changes. Optic disc changes were focal notching, optic disc haemorrhage, retinal nerve fiber layer (RNFL)defects, overpass-blood vessel crossing over an area of neuroretinal rim loss.Visual fields changes were the glaucoma hemifield test outside normal limits or a cluster of three or more non-edge points in a typical location of glaucoma or a corrected pattern standard deviation that occurs in less than 5% of normal visual fields

Exclusion Criteria:

* Exclusion criteria included history of uveitis or CME, substantial ocular irritation at baseline, or a history of intraocular surgery or a laser procedure within 6 months of baseline, the presence of systemic disorders that could be associated with uveitis or CME (ie, diabetes mellitus and rheumatologic diseases), presence of age-related macular degeneration and other macular diseases, pregnancy, breastfeeding, and inadequate contraception (in females), treatment with systemic beta-blocker, history of bronchial asthma, chronic obstructive pulmonary disease , sinus bradycardia, second and third degree atrioventricular block , sinoatrial block and functionally significant visual field loss

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change of mean flare values from baseline at 6 months | Flare measurements occurred at baseline; after 15 days; and after 1, 2, 3, 4, 5, and 6 months of treatment
  A flare measure of a laser flare meter (FM 500; Kowa Co Ltd, Tokyo, Japan) was used to determine the status of the blood-aqueous barrier at all follow-up visits. According to information provided by the manufacturer, flare readings greater than 26 photon counts per millisecond (p/ms) are indicative of a disruption in the blood-aqueous barrier.

SECONDARY OUTCOMES:
Change of mean macular thickness values from baseline at 6 months | Macular optical coherence tomography images were taken at baseline, after one month and six months of treatment, or if a patient has reduced visual acuity during follow-up
  Foveal macular thickness wiht Spectral Domain Optical Coherence Tomography (Cirrus Model 4000; Carl Zeiss Meditec, Dublin, California, USA) examination was conducted to investigate the occurrence of cystoid macular edema (CME). If CME was detected, the patient was instructed to discontinue taking the medication and a nonsteroidal anti-inflammatory drug was prescribed.

CONTACTS AND LOCATIONS:
Overall Officials: Alana M Santana, MD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- Hospital de Clínicas, UNICAMP, Campinas, São Paulo, Brazil